CLINICAL TRIAL: NCT00278707
Title: Phase 1 Treatment With GTA in Two Infant With Canavan Disease
Brief Title: GTA-Glyceryltriacetate for Canavan Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-05-3968-YA-CTIL
Record Dates: First submitted 2006-01-15; First posted 2006-01-18 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-08

CONDITIONS: Infantile Canavan Disease; Deficiency Disease, Aspartoacylase
Keywords: Canavan Disease; Aspartoacylase Deficiency; NAA; Acetate; Glyceryltriacetate
MeSH Terms: conditions — Canavan Disease

INTERVENTIONS:
Drug: GTA: Glyceryltriacetate

SUMMARY:
The purpose of this study is to determine whether oral supplementation of glyceryl triacetate improves the clinical prognosis of Canavan Disease.

DETAILED DESCRIPTION:
Canavan Disease is caused by a deficiency in the enzyme named Aspartoacylase (ASPA). This disease is a devastating, progressive disease with no available treatment. As a result of the ASPA deficiency, there are high levels of N-acetylaspartate (NAA) and low levels of L-aspartate and acetate.

We hypothesize that one of the functions of ASPA is to provide sufficient levels of acetate for CNS myelinization. For this reason, we offer to supplement acetate levels by the oral administration of glyceryl triacetate (GTA). Such treatment must be offered to patients before the age of 18 months, prior to the termination of CNS myelinization.

1. Two patients, aged less than 15 months, will receive daily doses of oral GTA
2. The daily dose will be increased incrementally until the maintenance dose is reached. This will be done under close monitoring of the patients, including periodic blood gas sampling.
3. GTA has not been shown to cause any known toxicity, according to the Cosmetic Ingredient Review Expert Panel (Fiume, 2003).

ELIGIBILITY:
Inclusion Criteria:

* Age below 15 months
* Biochemically diagnosed with Canavan Disease

Exclusion Criteria:

* None

Ages: 0 Years to 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5
Dates: Start 2006-01; Study Completion 2006-07

PRIMARY OUTCOMES:
All primary outcome will be evaluated 4 months following the initiation of treatment:
Neurological Status
Brain Imaging: MRI & MRS
NAA Levels in Urine
Ophthalmologic Examination

CONTACTS AND LOCATIONS:
Overall Officials: Yair Anikster, MD PI, Principal Investigator — Director Metabolic Disease Unit
Locations (1):
- Dr. Y. Anikster, Tel Aviv, Israel

REFERENCES:
- [Background] Mathew R, Arun P, Madhavarao CN, Moffett JR, Namboodiri MA. Progress toward acetate supplementation therapy for Canavan disease: glyceryl triacetate administration increases acetate, but not N-acetylaspartate, levels in brain. J Pharmacol Exp Ther. 2005 Oct;315(1):297-303. doi: 10.1124/jpet.105.087536. Epub 2005 Jul 7. PMID 16002461
- [Background] Madhavarao CN, Arun P, Moffett JR, Szucs S, Surendran S, Matalon R, Garbern J, Hristova D, Johnson A, Jiang W, Namboodiri MA. Defective N-acetylaspartate catabolism reduces brain acetate levels and myelin lipid synthesis in Canavan's disease. Proc Natl Acad Sci U S A. 2005 Apr 5;102(14):5221-6. doi: 10.1073/pnas.0409184102. Epub 2005 Mar 22. PMID 15784740